CLINICAL TRIAL: NCT01759706
Title: Safety and Feasibility Study of an Enhanced Recovery After Surgery Protocol in Patients Undergoing Elective Pancreaticoduodenectomy.
Brief Title: Safety and Feasibility Study of Enhanced Recovery in Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Braga, Professor in Surgery, Università Vita-Salute San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS_PANCREAS 01
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ondansetron; Dexamethasone; Calcium Dobesilate; Analgesia, Epidural; Ropivacaine; Sufentanil; Diazepam; sodium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Recovery After Surgery (ERAS) (Experimental): Patients treated with enhanced recovery after surgery protocol: preadmission counselling, preoperative immunonutrition, no preoperative bowel preparation, epidural analgesia with naropin + sufentanil, no pre-anesthetic medication, intraoperative iv fluid restriction, PONV prophylaxis with ondansetron + dexamethasone, hypothermia prophylaxis, removal of nasogastric tube (NGT) at the end of surgery, postoperative mobilization program, solid food diet from POD 2, early stop of iv infusions and removal of urinary catheter.
  Interventions: Behavioral: Enhanced recovery after surgery protocol; Drug: PONV prophylaxis with Ondansetron + Dexamethasone; Other: Postoperative mobilization program; Drug: Epidural analgesia with naropin + sufentanil; Behavioral: Preadmission counselling
- Standard perioperative care (Control) (Active Comparator): Patients treated with standard care perioperative protocol: epidural analgesia with naropin + sufentanil, pre-anesthetic medication with diazepam, Preoperative bowel preparation with sodium phosphate, removal of nasogastric tube on POD 1, solid food diet from POD 4
  Interventions: Procedure: Standard perioperative care; Drug: Epidural analgesia with naropin + sufentanil; Drug: Pre-anesthetic medication with diazepam; Drug: Preoperative bowel preparation with sodium phosphate

INTERVENTIONS:
Behavioral: Enhanced recovery after surgery protocol — ERAS items implemented were: preadmission counselling, preoperative immunonutrition, no preoperative bowel preparation, epidural analgesia, no pre-anesthetic medication, intraoperative iv fluid restriction, PONV and hypothermia prophylaxis, removal of nasogastric tube (NGT) at the end of surgery, mobilization protocol, solid food diet from POD 2, early stop of iv infusions and removal of urinary catheter.
  Arms: Enhanced Recovery After Surgery (ERAS)
Procedure: Standard perioperative care — Epidural analgesia, pre-anesthetic medication with diazepam, bowel preparation with oral assumption of sodium phosphate, removal of nasogastric tube on POD 1, solid food diet from POD 4
  Arms: Standard perioperative care (Control)
Drug: PONV prophylaxis with Ondansetron + Dexamethasone — Postoperative nausea and vomiting prophylaxis with Ondansetron + Dexamethasone.
  Other Names: Zofran + Decadron
  Arms: Enhanced Recovery After Surgery (ERAS)
Other: Postoperative mobilization program — Patient mobilization for 2 hours on first postoperative day Patient mobilization for 4 hours on first postoperative day + assisted deambulation in the room Patient mobilization for 6 hours on first postoperative day + assisted deambulation in the ward
  Arms: Enhanced Recovery After Surgery (ERAS)
Drug: Epidural analgesia with naropin + sufentanil — Midthoracic epidural analgesia with naropin 0.2 % plus sufentanil 0,5 mcg/mL
  Other Names: Disufen
Drug: Pre-anesthetic medication with diazepam — Premedication before general anesthesia
  Other Names: Valium
  Arms: Standard perioperative care (Control)
Behavioral: Preadmission counselling — Patient multidisciplinary preoperative counselling, including anesthesiologist, surgeon and nurse.
  Arms: Enhanced Recovery After Surgery (ERAS)
Drug: Preoperative bowel preparation with sodium phosphate — Preoperative bowel preparation with oral assumption of sodium phosphate
  Other Names: Phospho-Lax
  Arms: Standard perioperative care (Control)

SUMMARY:
The purpose of this study is to assess the adherence to an enhanced recovery after surgery (ERAS) pathway and the impact of the ERAS protocol on postoperative short-term outcome in patients undergoing pancreaticoduodenectomy (PD).

DETAILED DESCRIPTION:
A specific enhanced recovery after surgery (ERAS) protocol has been applied since October 2010 in consecutive patients undergoing pancreaticoduodenectomy (PD) in a high volume Institution. Patient compliance for each item has been assessed. Each ERAS patient was matched with a patient who received standard perioperative care. Match criteria were age, gender, malignant / benign disease, and PD prognostic score.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective pancreaticoduodenectomy

Exclusion Criteria:

* Intraoperative detection of metastatic disease (non-operability)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adherence to the pathway | Participants will be followed from two weeks before surgery, for the duration of hospital stay, and for 30 days after discharge, an expected average of 8 weeks.
  Adherence to single items of the pathway.

SECONDARY OUTCOMES:
Postoperative outcome | The outcomes will be assessed for the duration of hospital stay and for 30 days after discharge
  Comparison of postoperative morbidity and mortality, length of hospital stay, readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, MI, Italy

REFERENCES:
- [Background] Balzano G, Zerbi A, Braga M, Rocchetti S, Beneduce AA, Di Carlo V. Fast-track recovery programme after pancreatico- duodenectomy reduces delayed gastric emptying. Br J Surg. 2008 Nov;95(11):1387-93. doi: 10.1002/bjs.6324. PMID 18844251
- [Background] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. World J Surg. 2013 Feb;37(2):240-58. doi: 10.1007/s00268-012-1771-1. No abstract available. PMID 22956014